CLINICAL TRIAL: NCT07040319
Title: Phase I/II Study of the Pharmacokinetics and Safety of Glecaprevir/Pibrentasvir Initiated in Pregnancy in Women With Hepatitis C With and Without HIV
Brief Title: Study of the Pharmacokinetics and Safety of Glecaprevir/Pibrentasvir Initiated in Pregnancy in Women With Hepatitis C With and Without HIV
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT 2041
Record Dates: First submitted 2025-06-13; First posted 2025-06-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-06

CONDITIONS: Hepatitis C
Keywords: HIV; Hepatitis C; Pregnancy; Glecaprevir/Pibrentasvir
MeSH Terms: conditions — Hepatitis C | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GLE/PIB (Experimental): Pregnant participants will take three (3) GLE/PIB fixed-dose combination tablets orally once daily with food for eight weeks
  Interventions: Drug: Glecaprevir/pibrentasvir

INTERVENTIONS:
Drug: Glecaprevir/pibrentasvir — 100 mg glecaprevir and 40 mg pibrentasvir for a total daily dose of glecaprevir 300 mg/pibrentasvir 120 mg
  Other Names: GLE/PIB

SUMMARY:
This is a Phase I/II, multi-site, open-label, single arm study to describe the pharmacokinetics (PK) and safety of glecaprevir/pibrentasvir (GLE/PIB) initiated during pregnancy in women with hepatitis C virus (HCV) infection (acute or chronic) with or without HIV and to evaluate safety for their infants through 10 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Of legal age or circumstance to provide independent informed consent as determined by site standard operating procedures (SOPs) and consistent with institutional review board/ethics committee (IRB/EC) policies and procedures
* Willing and able to provide written informed consent for their own and their infant's study participation
* At entry, 16-45 years of age (inclusive)
* At entry, gestational age of 14-32 weeks, defined as greater than 13 weeks plus six days and less than or equal to 32 completed weeks gestation, as determined by the site investigator based on best obstetric estimate
* At screening and at study entry, no evidence of multiple gestation, fetal anomalies, or intrauterine fetal growth restriction, as determined by the site investigator based on ultrasound
* At screening, detectable HCV RNA test result based on testing of a specimen collected within 30 days prior to entry
* At screening, negative test results for hepatitis B surface antigen based on testing of a specimen collected within 30 days prior to entry
* At screening (i.e., from specimens collected within 30 days prior to entry), has normal, grade 1, grade 2, or grade 3 results for the following

  * Aspartate aminotransferase (AST) (<10.0 x ULN)
  * Alanine aminotransferase (ALT) (<10.0 x ULN)
* At screening (i.e., from specimens collected within 30 days prior to entry), has normal, grade 1, or grade 2 results for the following

  * Hemoglobin (≥8.5 g/dL)
  * Creatinine (≤1.8 x ULN)
* At screening (i.e., from specimens collected within 30 days prior to entry), has normal or grade 1 results for the following

  * International normalized ratio (INR) (<1.5 x ULN)
  * Platelet count (≥100,000 cells/mm3)
  * Total bilirubin (<1.6 x ULN)
* HIV status determined based on testing meeting the requirements specified in protocol
* For pregnant participants living with HIV: has a suppressed HIV viral load (HIV-1 RNA below the limit of quantification of the assay) on an ARV regimen for at least 30 consecutive days prior to entry that does not include efavirenz, etravirine, cobicistat, or any protease inhibitor (e.g., atazanavir, darunavir, lopinavir, ritonavir), as determined by the site investigator based on available medical records
* At entry, expects to remain in the geographic area of the study site during pregnancy and for 10 weeks postpartum (or for 20 weeks post-entry, depending on gestational age at entry), as determined by the site investigator based on pregnant participant report

Exclusion Criteria:

* Any previous treatment for hepatitis C, including HCV DAAs or interferon-based treatment
* High risk of preterm delivery, defined as either of the following:

  * History of spontaneous preterm delivery at less than 34 weeks, as determined by the site investigator based on pregnant participant report and available medical records, or
  * Shortened cervix less than 20 mm if noted on ultrasound during the current pregnancy, as determined by the site investigator based on available medical records
* Receipt of any prohibited medication, within 14 days prior to entry, as determined by the site investigator based on pregnant participant report and available medical records
* Any of the following liver-related conditions:

  * Clinical diagnosis of acute hepatitis not otherwise attributable to hepatitis C with AST or ALT ≥2.5 x ULN
  * Evidence of decompensated cirrhosis including history of or present variceal hemorrhage, ascites, spontaneous bacterial peritonitis, hepatic encephalopathy, hepatocellular carcinoma, hepatorenal syndrome, or hepatopulmonary syndrome
* Has any other documented or suspected clinically significant medical condition or any other condition that, in the opinion of the site investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Geometric mean AUC0-24h | At weeks 3 & 6
  Area under the curve from start of dose to 24 hours post dose
Geometric mean Cmax | At weeks 3 & 6
  Peak concentration from start of dose to 24 hours post dose
Geometric mean C24h | At weeks 3 & 6
  Concentration at 24 hours post dose
Percentage of pregnant/ postpartum participants who experience a grade 3 or higher adverse event assessed as related to study drug | Initiation of treatment to a) completion of treatment and b) latter of 10 weeks post-partum or 20 weeks post treatment initiation
Percentage of pregnant participants who experience a serious adverse event assessed as related to study drug | Initiation of treatment to a) completion of treatment and b) latter of 10 weeks post-partum or 20 weeks post treatment initiation

SECONDARY OUTCOMES:
Percentage of pregnant/postpartum participants with sustained virologic response (SVR12) | 12 weeks after planned treatment completion
  defined as unquantifiable hepatitis C RNA (less than the lower limit of quantification [<LLOQ])
Percentage of pregnant participants with spontaneous abortions or miscarriage | At birth/delivery
  (<20 weeks gestation)
Percentage of pregnant participants with stillbirths | At birth/delivery
  (≥20 weeks gestation)
Percentage of infants small for gestational age | At birth/delivery
  <10th percentile
Percentage of infants with low birth weight | At birth/delivery
  <2500 g
Percentage of pre-term births | At birth/delivery
  <37 weeks gestation
Percentage of pregnancies with occurrence of any of the following adverse pregnancy events | At birth/delivery
  spontaneous abortion or miscarriage, stillbirth, small gestational age, low birth weight, or preterm birth
Percentage of infants with a congenital abnormality | At birth/delivery
Percentage of infants with a grade 5 adverse event | From birth through 10 weeks of age
Percentage of infants with Grade 3 or higher adverse event assessed as related to study drug | From birth through 10 weeks of age
Percentage of infants with a serious adverse events assessed as related to study drug | From birth through 10 weeks of age
Percentage of occurrence of any of the following in infants: grade 5 adverse event within 28 days of birth, grade 3 or higher adverse event assessed as related to study drug, or severe adverse event assessed as related to study drug | From birth through 10 weeks of age
Median weight of infants | At birth and 10 weeks of age
Median length of infants | At birth and 10 weeks of age
Median head circumference of infants | At birth and 10 weeks of age
Percentage of infants with quantifiable hepatitis C RNA | At 10 or more weeks of age

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - USC LA, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of Colorado Denver, Aurora, Colorado
  - Univ. of Florida Jacksonville, Jacksonville, Florida
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins University Baltimore, Baltimore, Maryland
  - SUNY Stony Brook, Stony Brook, New York
  - Bronx-Lebanon Hospital Center, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - Baylor College of Medicine//Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: * Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses?
  * To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available?
  * Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https:// www.impaactnetwork.org/ resources/study-proposals.htm. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.